CLINICAL TRIAL: NCT03613194
Title: Mechanistic and Molecular Study of the Process of Metastatic Dissemination in Colorectal Cancer
Acronym: DISCOVER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-A02878-45; 2017/2511 (Other: CSET number)
Record Dates: First submitted 2018-07-19; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with metastatic colorectal cancer (Other): After inclusion in the study, eligible patients having hepatic metastases and/or péritonéales of a colorectal cancer considered as resecables will have biological and tissue samples.
  The samples will be carried out at the time of the surgical gesture envisaged under general anaesthesia and will concern:
  * Tumoral material: primitive tumour (if available), hepatic metastases and/or peritoneal
  * Peritoneal liquid
  * none tumoral peritoneum
  * Portal blood
  * Peripheral blood
  * Cellulo-lymphatic material The necessary time to carry out the whole of these samples is estimated at 10-15 minutes maximum.
  In the event of complex situations being able to complicate the surgical gesture initially envisaged or to increase by them morbidity, one or more these samples will not be carried out. This decision will be made at the discretion of the investigator.
  Interventions: Procedure: Sampling

INTERVENTIONS:
Procedure: Sampling — After inclusion in the study, eligible patients having hepatic metastases and/or péritonéales of a colorectal cancer considered as resecables will have biological and tissue samples.
  The samples will be carried out at the time of the surgical gesture envisaged under general anaesthesia and will concern:
  * Tumoral material: primitive tumour (if available), hepatic metastases and/or peritoneal
  * Peritoneal liquid
  * none tumoral peritoneum
  * Portal blood
  * Peripheral blood
  * Cellulo-lymphatic material The necessary time to carry out the whole of these samples is estimated at 10-15 minutes maximum.
  In the event of complex situations being able to complicate the surgical gesture initially envisaged or to increase by them morbidity, one or more these samples will not be carried out. This decision will be made at the discretion of the investigator.

SUMMARY:
To confirm the role of the collective dissemination in the mechanisms of tumoral invasion of colorectal cancers

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Histological Diagnosis of stage IV colorectal cancer
* Hepatic metastasis and/or peritoneal potentially resecable
* Patient affiliated with a mode of the social security or recipient of such a mode
* Information of the patient or his legal representative and collection of his assent

Exclusion Criteria:

* None metastatic colorectal cancer
* Cancer of appendicular origin
* Patients deprived of liberty or unable to give his assent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06-25 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Identification and characterization of the tumoral intermediaries on the overflowing peritoneal | Up to 24 months
  After several separation and centrifugation steps, clusters and tumor cells are isolated and counted in the various biological samples. The different isolated intermediates will be analyzed by immunolabeling with the antibodies directed against CK20, EpCAM, Vimentine and CD45.
Identification and characterization of the tumoral intermediaries on the portal blood | Up to 24 months
  After several separation and centrifugation steps, clusters and tumor cells are isolated and counted in the various biological samples. The different isolated intermediates will be analyzed by immunolabeling with the antibodies directed against CK20, EpCAM, Vimentine and CD45.
Identification and characterization of the tumoral intermediaries on the peripheral blood | Up to 24 months
  After several separation and centrifugation steps, clusters and tumor cells are isolated and counted in the various biological samples. The different isolated intermediates will be analyzed by immunolabeling with the antibodies directed against CK20, EpCAM, Vimentine and CD45.
Identification and characterization of the tumoral intermediaries on the hepatic metastasis and/or peritoneal) | Up to 24 months
  After several separation and centrifugation steps, clusters and tumor cells are isolated and counted in the various biological samples. The different isolated intermediates will be analyzed by immunolabeling with the antibodies directed against CK20, EpCAM, Vimentine and CD45.

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No